CLINICAL TRIAL: NCT02620293
Title: A 47 Hour, Single Application, Occlusive Forearm Skin Patch Test to Assess, Under Dermatological Control, the Acute Cutaneous Tolerance of Project Storm on the Forearm of Adult Subjects With Dry/Atopic and Very Dry/Atopic Skin
Brief Title: A 47 Hour Occlusive Cutaneous Skin Patch Test on Adult Subjects With Dry/Atopic Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Skin Investigation Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 09224-01
Record Dates: First submitted 2015-09-09; First posted 2015-12-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eczema Emollient (Experimental): Eczema Repair Emollient
  Interventions: Device: Eczema Repair Emollient

INTERVENTIONS:
Device: Eczema Repair Emollient — An Emollient

SUMMARY:
This is an open label, non-comparative investigation to determine the tolerance of Eczema Repair Emollient on healthy subjects with dry/atopic and very dry/atopic skin.

The Eczema Repair Emollient will be applied for 47 hours under occlusion. Skin tolerance will be assessed immediately and 1 hour, 24, 48 and 72 hours after patch removal.

DETAILED DESCRIPTION:
At immediate, 1, 24, 48, and 72 hours post-test patch removal (date & time of each assessment will be recorded), each test site will be scored for erythema and oedema by the trained investigator using the ISO 10993 scoring system.

Primary Endpoint The irritation of the test product according to the Cutaneous Irritancy Index value. The test product should be graded as 'non-irritant' and confirmed by the study dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give written informed consent and from whom written informed consent has been obtained
* Generally healthy male and female subjects between the ages of 18 and 65 years inclusive
* Subjects assessed by the dermatologist as having dry/atopic and very dry/ atopic skin
* Subjects who are able to understand the study, co-operate with the study procedures and are able to attend for all study assessments

Exclusion Criteria:

* Subjects with active Psoriasis or other active skin disorders or with present skin tumours or malignant disease or a history of those
* Subjects taking antihistamine or corticoids, any medication for the treatment of diabetes mellitus, immuno-suppressive drugs or any other medication which in the opinion of the dermatologist may affect the test results.
* Subjects with active skin disorders or a history of skin disorders (e.g. psoriasis, eczema, vitiligo, pityriasis versicolor, acne) which in the opinion of the trainee dermatologist or SIT personnel may affect the test results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Skin tolerance assessment using the ISO 10993 scoring system through visual assessment | 47 hours
  Irritation of test products assessed using the Cutaneous Irritancy Index (scores range from <1 which is non-irritant to >4 strongly irritating

CONTACTS AND LOCATIONS:
Overall Officials: Dörte Segger, PhD, Principal Investigator — Skin Investigational Technology
Locations (1):
- Skin Investigation Technology, Hamburg, Germany